CLINICAL TRIAL: NCT06329921
Title: Inpatient Monitoring of Unfractionated Heparin
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Tillman, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 232192
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Blood Clot; Thrombosis
Keywords: heparin; anticoagulation; anti-Xa; PTT
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic, randomized controlled clinical trial with parallel group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: PTT protocol (Active Comparator): Patients randomized to this arm will be monitored using the nurse-managed PTT guided protocol. This includes patients on both high- and low-dose heparin protocols.
  Interventions: Other: PTT protocol
- Active Comparator: anti-Xa protocol (Active Comparator): Patients randomized to this arm will be monitored using the pharmacy-managed anti-Xa protocol. This includes patients on both high- and low-dose heparin protocols.
  Interventions: Other: anti-Xa protocol

INTERVENTIONS:
Other: PTT protocol — Patients will be monitored using the nurse-managed PTT protocol.
  Arms: Active Comparator: PTT protocol
Other: anti-Xa protocol — Patients will be monitored using the pharmacy-managed anti-Xa protocol.
  Arms: Active Comparator: anti-Xa protocol

SUMMARY:
Unfractionated heparin (UFH) is the most widely used intravenous (IV) anticoagulant for treating and preventing thromboembolic disease (e.g., blood clots ). UFH must be closely monitored and adjusted in the hospital. There are two assays used to monitor UFH: 1) the activated partial thromboplastin time (PTT) and 2) the chromogenic anti-factor Xa assay (anti-Xa). This study aims to compare PTT and anti-Xa methods for monitoring UFH in a pragmatic, randomized controlled trial to determine which helps patients reach a therapeutic anticoagulation range faster.

DETAILED DESCRIPTION:
Unfractionated heparin (UFH) is the most widely used intravenous (IV) anticoagulant for the treatment and prevention of thromboembolic disease (e.g., blood clots ). When administered by intravenous injection, the onset of action is immediate. Indications for use of UFH include venous thromboembolism, acute coronary syndrome, and acute ischemic stroke. UFH is used to prevent thrombosis in the setting of arrhythmias, extracorporeal membrane oxygenation (ECMO), cardiopulmonary bypass (CPB), and endovascular procedures. The unpredictable pharmacokinetics of UFH and interpatient variability result in a narrow therapeutic index restricting its use to the hospital setting with close monitoring and adjustments.

Two validated assays exist and are in use at the VUMC adult hospital for the monitoring of unfractionated heparin: 1) the activated partial thromboplastin time (PTT) and 2) the chromogenic anti-factor Xa assay (anti-Xa). At VUMC, the PTT protocol is managed by nursing; the anti-Xa protocol is managed by clinical pharmacy. Both are clinically acceptable methods for titration and adjustment of unfractionated heparin. Assessing the therapeutic effect of unfractionated heparin is most often performed with the PTT, which requires institutional calibration to a specific heparin level to account for the variable PTT responses with different commercial reagents and laboratory instruments. The PTT can be influenced by various elements during sample processing, laboratory analysis, and patient biological factors that may cause it to be an inaccurate indication of the degree of anticoagulation. This can lead to patients not getting the correct heparin dosing for their clinical needs.

The anti-Xa assay is another method of measuring the degree of therapeutic effect of heparin. In routine clinical practice the anti-Xa is not as widely available and less familiar among many providers. This assay can be impacted by variability in sample collection and processing and laboratory analysis. Compared to the PTT assay, however, it is much less influenced by patient-specific biological factors. This may help improve heparin monitoring and titration to ensure patients receive therapeutic levels of anticoagulation and do not get too much or too little heparin. However, large studies using anti-Xa for management of heparin in the treatment of venous thromboembolism have not been performed.

PTT and anti-Xa heparin monitoring protocols have not been compared in a prospective, randomized setting. The study team will conduct a pragmatic, randomized clinical trial comparing the effectiveness of both methods for optimal monitoring of intravenous unfractionated heparin for systemic anticoagulation in hospitalized adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Vanderbilt University Hospital age 18 years and older who are admitted as observation or inpatients for whom intravenous unfractionated heparin (monitored via the PTT nurse-managed protocol) is ordered.
* Baseline PTT value is ≥0 and ≤ 36.0 seconds
* Baseline heparin level anti-Xa assay value is ≥0 and ≤0.3

Exclusion Criteria:

* Indication for anticoagulation is extracorporeal membrane oxygenation or cerebrovascular ischemic event.
* Provider determines patient is not appropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time to therapeutic anticoagulation range | Randomization to hospital discharge at approximately 5-7 days post-randomization
  Time to reach therapeutic anticoagulation range by coagulation assay

SECONDARY OUTCOMES:
Measurements in therapeutic anticoagulation range | Randomization to hospital discharge at approximately 5-7 days post-randomization
  Percent of measurements in therapeutic range per coagulation assay, as defined by assay protocol
Coagulation laboratory measurements | Randomization to hospital discharge at approximately 5-7 days post-randomization
  The number of coagulation laboratory measurements for overall in-hospital coagulation time.
New thrombotic events | Randomization to hospital discharge at approximately 5-7 days post-randomization and for 24 hours after anticoagulation cessation.
  Incidence of new thrombotic events on anticoagulation and within 24 hours of anticoagulation cessation
New clinically relevant bleeding events | Randomization to 48 hours after anticoagulation cessation, approximately 5-7 days post-randomization
  Incidence of clinically relevant bleeding adverse events (overt events or decline in hemoglobin >2 g/dL over a 24-hour period, or leading to transfusion of two or more units of whole blood or red blood cells, within 48 hours of anticoagulation cessation)
New coagulation events | Randomization to 48 hours after anticoagulation cessation, approximately 5-7 days post-randomization
  Incidence of new coagulation events on anticoagulation, including thrombotic events and clinically relevant bleeding adverse events as defined in Outcomes 4 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tillman, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Hirsh J, Warkentin TE, Raschke R, Granger C, Ohman EM, Dalen JE. Heparin and low-molecular-weight heparin: mechanisms of action, pharmacokinetics, dosing considerations, monitoring, efficacy, and safety. Chest. 1998 Nov;114(5 Suppl):489S-510S. doi: 10.1378/chest.114.5_supplement.489s. No abstract available. PMID 9822059
- [Background] Smythe MA, Priziola J, Dobesh PP, Wirth D, Cuker A, Wittkowsky AK. Guidance for the practical management of the heparin anticoagulants in the treatment of venous thromboembolism. J Thromb Thrombolysis. 2016 Jan;41(1):165-86. doi: 10.1007/s11239-015-1315-2. PMID 26780745
- [Background] Eikelboom JW, Hirsh J. Monitoring unfractionated heparin with the aPTT: time for a fresh look. Thromb Haemost. 2006 Nov;96(5):547-52. PMID 17080209
- [Background] Olson JD, Arkin CF, Brandt JT, Cunningham MT, Giles A, Koepke JA, Witte DL. College of American Pathologists Conference XXXI on laboratory monitoring of anticoagulant therapy: laboratory monitoring of unfractionated heparin therapy. Arch Pathol Lab Med. 1998 Sep;122(9):782-98. PMID 9740136
- [Background] Wool GD, Lu CM; Education Committee of the Academy of Clinical Laboratory Physicians and Scientists. Pathology consultation on anticoagulation monitoring: factor X-related assays. Am J Clin Pathol. 2013 Nov;140(5):623-34. doi: 10.1309/AJCPR3JTOK7NKDBJ. PMID 24124140
- [Background] Marlar RA, Clement B, Gausman J. Activated Partial Thromboplastin Time Monitoring of Unfractionated Heparin Therapy: Issues and Recommendations. Semin Thromb Hemost. 2017 Apr;43(3):253-260. doi: 10.1055/s-0036-1581128. Epub 2016 Jun 6. PMID 27272964

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT06329921/SAP_001.pdf